CLINICAL TRIAL: NCT04365959
Title: Study of the Feasibility and Usefulness of the Prone Position in Patients With Respiratory Distress From Covid-19 Not Intubated, in Spontaneous Breath in Oxygen Therapy or Cpap
Brief Title: The Prone Position in Covid-19 Affected Patients
Acronym: PRON-COVID
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: PRON-COVID
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Sars-CoV2
Keywords: COVID-19; sars-covid-2
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid-19 pneumonia related patients: This study will be conducted on all patients admitted to the Infectious Diseases and UTIR units of the S. Gerardo Hospital in Monza with the diagnosis of related COVID pneumonia requiring oxygen support or CPAP.
  Interventions: Procedure: Prone position

INTERVENTIONS:
Procedure: Prone position — The objective of the study is to value the ability of the prone position to increase the oxygenation of the patient with SARS-cov-2 pneumonia as a lung recruitment index; the PP also prevents the need for intubation and the consequent risk deriving from the procedure itself and from the predisposition to develop superinfections (VAP).
  Other Names: PP

SUMMARY:
The prone position during mechanical ventilation in patients with Acute Respiratory Distress Syndrome (ARDS) is able to improve oxygenation and thus reduce mortality. The objective of the study is to evaluate the ability of the prone position to increase the oxygenation of the patient with SARS-cov-2 pneumonia.

DETAILED DESCRIPTION:
BACKGROUND:

It has been shown that the prone position (PP) during mechanical ventilation (VM) in patients with Acute Respiratory Distress Syndrome (ARDS) is able to improve oxygenation and thus reduce mortality.

The reduced mortality, however, is not only caused by an increase in oxygen, but also by the ability of the PP to reduce the damage associated with mechanical ventilation (VILI).

Studies show that the benefits of PP are also present in non-intubated patients; the PP prevents the need for intubation and the consequent risk deriving from the procedure itself and from the predisposition to develop superinfections (VAP).

Moreover, a reduction in the need for intubation and therefore hospitalization in the ICU would be particularly useful in a context of great health emergency with limited resources.

The objective of the study is to value the ability of the prone position to increase the oxygenation of the patient with SARS-cov-2 pneumonia as a lung recruitment index.

STUDY DESIGN:

This is a monocentric study that will be conducted on all patients admitted to the Infectious Diseases and UTIR units of the S. Gerardo Hospital in Monza with the diagnosis of related COVID pneumonia requiring oxygen support or CPAP.

Sample size (n. Patients): 56

The duration of enrollment is estimated in 1 month. Patients will be monitored until discharged from the hospital. The overall duration of the study is estimated to be 1 year (including enrollment, follow up and data analysis).

The patient will be enrolled in the study when consent is obtained. The following data will be collected:

* Patient registration
* Demographic and anthropometric data
* Comorbidity and lifestyle habits
* Hospitalization data
* Blood chemistry tests
* Ventilation parameters

After 10 minutes and at the end of pronation, the feasibility of pronation and ventilation parameters will also be assessed.

STATISTICAL ANALYSIS:

Clinical data relating to enrolled patients will be analysed by means of descriptive statistics on continuous quantitative variables using indicators chosen on the basis of the distributional form. Categorical variables will be described in percentages. Hypotheses on PaO2 / FiO2 performance will be verified through the T test for paired data if the distributional form allows it or alternatively the Wilcoxon test will be used. In this case we will proceed with a recalculation of the power study.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years old or <= 75 years old
* Diagnosis of COVID related pneumonia requiring oxygen or CPAP support

Exclusion Criteria:

* pregnant patients
* patients with impaired consciousness and / or uncooperative
* patients with NYHA class> II
* patients with high proBNP
* patients with COPD
* contraindications evidenced by the physicians

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on all patients admitted to the Infectious Diseases and UTIR units of the S. Gerardo Hospital in Monza with the diagnosis of related COVID pneumonia requiring oxygen or CPAP support.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Number of patients in whom the prone position caused an increase in oxygenation | Until patient discharge from the hospital (approximately 1 month after enrollment)
  Measure the ability of the prone position to increase the oxygenation of the patient with SARS-cov-2 pneumonia as a lung recruitment index.

SECONDARY OUTCOMES:
The feasibility of prone position | Until patient discharge from the hospital (approximately 1 month after enrollment)
  Measure the feasibility of the prone position in terms of patient comfort and health resources in a context of a national health emergency.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Foti, Prof., Principal Investigator — ASST Monza-University Milano Bicocca
Locations (1):
- ASST Monza, Monza, MB, Italy

REFERENCES:
- [Background] Bouadma L, Lescure FX, Lucet JC, Yazdanpanah Y, Timsit JF. Severe SARS-CoV-2 infections: practical considerations and management strategy for intensivists. Intensive Care Med. 2020 Apr;46(4):579-582. doi: 10.1007/s00134-020-05967-x. Epub 2020 Feb 26. No abstract available. PMID 32103284
- [Background] Pappert D, Rossaint R, Slama K, Gruning T, Falke KJ. Influence of positioning on ventilation-perfusion relationships in severe adult respiratory distress syndrome. Chest. 1994 Nov;106(5):1511-6. doi: 10.1378/chest.106.5.1511. PMID 7956412
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Albert RK, Leasa D, Sanderson M, Robertson HT, Hlastala MP. The prone position improves arterial oxygenation and reduces shunt in oleic-acid-induced acute lung injury. Am Rev Respir Dis. 1987 Mar;135(3):628-33. doi: 10.1164/arrd.1987.135.3.628. PMID 3030168
- [Background] Hopkins SR, Henderson AC, Levin DL, Yamada K, Arai T, Buxton RB, Prisk GK. Vertical gradients in regional lung density and perfusion in the supine human lung: the Slinky effect. J Appl Physiol (1985). 2007 Jul;103(1):240-8. doi: 10.1152/japplphysiol.01289.2006. Epub 2007 Mar 29. PMID 17395757
- [Background] Mure M, Glenny RW, Domino KB, Hlastala MP. Pulmonary gas exchange improves in the prone position with abdominal distension. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1785-90. doi: 10.1164/ajrccm.157.6.9711104. PMID 9620906
- [Background] Albert RK, Hubmayr RD. The prone position eliminates compression of the lungs by the heart. Am J Respir Crit Care Med. 2000 May;161(5):1660-5. doi: 10.1164/ajrccm.161.5.9901037. PMID 10806172
- [Background] Broccard AF, Shapiro RS, Schmitz LL, Ravenscraft SA, Marini JJ. Influence of prone position on the extent and distribution of lung injury in a high tidal volume oleic acid model of acute respiratory distress syndrome. Crit Care Med. 1997 Jan;25(1):16-27. doi: 10.1097/00003246-199701000-00007. PMID 8989171
- [Background] Valenza F, Guglielmi M, Maffioletti M, Tedesco C, Maccagni P, Fossali T, Aletti G, Porro GA, Irace M, Carlesso E, Carboni N, Lazzerini M, Gattinoni L. Prone position delays the progression of ventilator-induced lung injury in rats: does lung strain distribution play a role? Crit Care Med. 2005 Feb;33(2):361-7. doi: 10.1097/01.ccm.0000150660.45376.7c. PMID 15699840
- [Background] Valter C, Christensen AM, Tollund C, Schonemann NK. Response to the prone position in spontaneously breathing patients with hypoxemic respiratory failure. Acta Anaesthesiol Scand. 2003 Apr;47(4):416-8. doi: 10.1034/j.1399-6576.2003.00088.x. PMID 12694139
- [Background] Scaravilli V, Grasselli G, Castagna L, Zanella A, Isgro S, Lucchini A, Patroniti N, Bellani G, Pesenti A. Prone positioning improves oxygenation in spontaneously breathing nonintubated patients with hypoxemic acute respiratory failure: A retrospective study. J Crit Care. 2015 Dec;30(6):1390-4. doi: 10.1016/j.jcrc.2015.07.008. Epub 2015 Jul 16. PMID 26271685
- [Derived] Coppo A, Bellani G, Winterton D, Di Pierro M, Soria A, Faverio P, Cairo M, Mori S, Messinesi G, Contro E, Bonfanti P, Benini A, Valsecchi MG, Antolini L, Foti G. Feasibility and physiological effects of prone positioning in non-intubated patients with acute respiratory failure due to COVID-19 (PRON-COVID): a prospective cohort study. Lancet Respir Med. 2020 Aug;8(8):765-774. doi: 10.1016/S2213-2600(20)30268-X. Epub 2020 Jun 19. PMID 32569585